CLINICAL TRIAL: NCT03386877
Title: Human Intrabony Defect Regeneration With Micro-grafts Containing Dental Pulp Stem Cells: a Randomized Controlled Clinical Trial.
Brief Title: Periodontal Regeneration Using Dental Pulp Stem Cells (DPSCs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Francesco Ferrarotti, Adjunct Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTurin stem cell RCT
Record Dates: First submitted 2017-12-15; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Guided Tissue Regeneration, Periodontal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental pulp stem cells (Experimental): Test sites (n=15) Periodontal regeneration using micro-grafts of Dental pulp stem cells seeded onto collagen sponge
  Interventions: Procedure: periodontal regeneration
- coagulum (Active Comparator): control sites (n=14) Periodontal regeneration using coagulum and collagen sponge alone
  Interventions: Procedure: periodontal regeneration

INTERVENTIONS:
Procedure: periodontal regeneration — Defects were accessed with the MIST In the test group the obtained micro-grafts enriched in DPSCs were endorsed onto a collagen sponge scaffold (Condress®, Istituto Gentili, Milano, Italy) to form a bio-complex. In the control group the collagen sponge was only hydrated using physiologic sterile solution. The collagen sponge with or without cells was provided to the masked surgeon who filled the intrabony defect. The flaps were repositioned and tension-free primary flap closure was obtained using horizontal internal mattress and interrupted sutures

SUMMARY:
The goal of this study is to evaluate if dental pulp stem cells (DPSCs) delivered into intrabony defects in a collagen scaffold would enhance the clinical and radiographic parameters of periodontal regeneration.

DETAILED DESCRIPTION:
In this randomized controlled trial, 29 chronic periodontitis patients presenting one deep intrabony defect and requiring extraction of one vital tooth were consecutively enrolled. Defects were randomly assigned to test or control treatments which both consisted of the use of minimally invasive surgical technique. The dental pulp of the extracted tooth was mechanically dissociated to obtain micro-grafts rich in autologous DPSCs. Test sites (n=15) were filled with micro-grafts seeded onto collagen sponge, whereas control sites (n=14) with collagen sponge alone. Clinical and radiographic parameters were recorded at baseline, 6 and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of advanced chronic periodontitis
* FMPS<20%
* FMBS<20%
* infrabony defect >2mm
* Probing depth >5mm
* presence of 1 vital and intact tooth requiring an extraction as autologous source of DPSCs

Exclusion Criteria:

* smoking
* controindicazion for periodontal surgery
* systemic diseases affecting periodontal healing
* pregnancy an lactation
* fixed orthodontic appliance
* history of periodontal surgery at the experimental teeth
* prostethic restorations at the experimental teeth
* furcation defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Radiographic bone fill | baseline and 12 months
  Periapical standardized radiographs were taken by a clinician masked to the clinical measurements using the paralleling technique and individually customized bite-blocks (RINN XCP Film Holding Instruments, Dentsply, York, USA)

SECONDARY OUTCOMES:
Probing depth reduction | baseline, 6 and 12 months
  Probing depth is assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)
Clinical attachment gain | baseline, 6 and 12 months
  Clinical attachment level is assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)
Recession reduction | baseline, 6 and 12 months
  Recession depth is assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Aimetti, Principal Investigator — Turin University
Locations (2):
- Italy (2):
  - CIR Dental school Turin University, Turin, Piedmont
  - CIR dental school, Turin, Piedmont